CLINICAL TRIAL: NCT06730802
Title: Protective Effect of PCSK9 Inhibitor Against Negative Inflammatory Response and Organ Dysfunction After Coronary Artery Bypass Grafting (PANDA VIII)
Acronym: PANDA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator of Department of Cardiovascular Surgery, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PANDA VIII
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Myocardial Ischaemic Syndrome; Coronary Heart Disease
Keywords: inflammation; CABG
MeSH Terms: conditions — Coronary Disease; Inflammation | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCSK9 inhibitor (Experimental): the experiment group will receive first PCSK9 inhibitor before CABG, then twice a month until 3 months later
  Interventions: Drug: PCSK9 inhibitor
- Statin (Sham Comparator): the control group will receive standard statin therapy.
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: PCSK9 inhibitor — the experiment group will receive first PCSK9 inhibitor before CABG, then twice a month until 3 months later.
  Arms: PCSK9 inhibitor
Drug: Statin — the control group will receive standard statin therapy.
  Arms: Statin

SUMMARY:
This is a multi-center, randomized controlled study to investigate whether early offering PCSK9 inhibitor can protect against negative inflammatory response and organ dysfunction after coronary artery bypass grafting (CABG). Subjects with myocardial ischaemic syndromes (MIS) will be enrolled in this study after consent information. After randomization, the control group will receive standard therapy, while the experiment group will receive first PCSK9 inhibitor before CABG, then twice a month until 3 months later. Six month after CABG, CRP will be used to evaluate inflammation, and echocardiography and coronary CTA will be used to evaluate cardiovascular function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Patients with myocardial ischemic syndromes (with any of the following):
* Patients are ready to undergo coronary artery bypass grafting (CABG) with 1 month;
* Participate voluntarily and sign an informed consent

Exclusion Criteria:

i. Pregnant and lactating women ii. During the study period and within 3 months of receiving the last dose of the study drug, women with fertility intentions and men unwilling to use effective contraceptive methods iii. Have used PCSK9 inhibitors within 3 months before enrollment, or have a history of severe allergic reactions to PCSK9 inhibitors iv. Severe infections requiring intravenous antibiotics v. HIV-positive or history of acquired immunodeficiency syndrome (AIDS) vi. With cognitive impairment or psychiatric illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular and Cerebrovascular Events | 6 months after surgery
  Major Adverse Cardiovascular and Cerebrovascular Events include cardiac death, reinfarction, emergency coronary revascularization and stroke

SECONDARY OUTCOMES:
C-reactive protein | 6 months after surgery
  Peripheral blood C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Lu-yao Ma, MD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (2):
- China (2):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oyama K, Furtado RHM, Fagundes A Jr, Zelniker TA, Tang M, Kuder J, Murphy SA, Hamer A, Wang H, Keech AC, Giugliano RP, Sabatine MS, Bergmark BA. Effect of Evolocumab on Complex Coronary Disease Requiring Revascularization. J Am Coll Cardiol. 2021 Jan 26;77(3):259-267. doi: 10.1016/j.jacc.2020.11.011. Epub 2020 Nov 13. PMID 33197560
- [Background] Na HR, Kwon OS, Kang JK, Kim YH, Lim JY. Evolocumab administration prior to Coronary Artery Bypass Grafting in patients with multivessel coronary artery disease (EVOCABG): study protocol for a randomized controlled clinical trial. Trials. 2022 May 23;23(1):430. doi: 10.1186/s13063-022-06398-3. PMID 35606883
- [Background] Nasso G, Larosa C, Bartolomucci F, Brigiani MS, Contegiacomo G, Demola MA, Vignaroli W, Tripoli A, Girasoli C, Lisco R, Trivigno M, Tunzi RM, Loizzo T, Hila D, Franchino R, Amodeo V, Ventra S, Diaferia G, Schinco G, Agro FE, Zingaro M, Rosa I, Lorusso R, Del Prete A, Santarpino G, Speziale G. Safety and Efficacy of PCSK9 Inhibitors in Patients with Acute Coronary Syndrome Who Underwent Coronary Artery Bypass Grafts: A Comparative Retrospective Analysis. J Clin Med. 2024 Feb 4;13(3):907. doi: 10.3390/jcm13030907. PMID 38337601